CLINICAL TRIAL: NCT01036217
Title: Evaluation of Potential Research Subjects - Screening Protocol for Clinical Studies
Brief Title: Screening Protocol for the Evaluation of Research Participants
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906412; 06-DA-N412
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-17

CONDITIONS: Substance Abuse; Disorders
Keywords: Recruitment; Adult; Telephone; Selection; Testing
MeSH Terms: conditions — Substance-Related Disorders; Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The National Institute on Drug Abuse (NIDA) uses a standardized set of procedures to develop a pool of potential participants for research studies. Because some of the data collected during screening are used later for research, the screening itself is considered a study. An applicant to any NIDA study is considered a participant in NIDA screening.

Objectives:

- To identify, recruit, and screen participants for NIDA research protocols.

Eligibility:

- Individuals 18 years of age and older who are able to provide informed consent.

Design:

* Individuals who are eligible for screening will undergo two interviews: a telephone interview and an in-person interview. The phone interview will determine eligibility for the in-person interview.
* The in-person interview may require up to five visits to NIDA. The in-person visit will involve any or all of the following procedures: (1) full physical examination and medical history; (2) psychiatric interview; (3) psychological testing; (4) electrocardiogram; (5) samples of blood, urine, and hair; and (6) other minimally invasive procedures as directed by the research staff.
* During screening, a photograph will be taken for confirmation of identity during subsequent visits for other studies.
* No clinical care will be provided as part of screening.

DETAILED DESCRIPTION:
Through its clinical research protocols, the NIDA IRP attempts to: elucidate the nature of drug abuse and addiction; determine the potential use of new therapies, both pharmacological and psychosocial; and decipher the long-term effects of drugs of abuse on the development, maturation, function, and structure of the brain and other organ systems. In support of the IRP's work, the scientific goal of this screening protocol is to assess potential research participants' eligibility for NIDA IRP research studies. Screening will include medical and psychological tests and procedures. The data collected during screening are a unique and valuable source of information that aids in NIDA's mission. Therefore, a secondary goal of this protocol is to obtain data that characterizes the population of subjects contacting NIDA about research participation and to analyze data so obtained, such as that on the prevalence and consequences of HIV/AIDS, viral hepatitis, and related diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults (at least age 18)
  2. Ability to understand and answer the questions as posed.

EXCLUSION CRITERIA:

1. Inability to provide valid informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55000 (Estimated)
Dates: Start 2006-05-17; Study Completion 2010-06-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States